CLINICAL TRIAL: NCT07058766
Title: Development of Post-Disaster Care Protocol for Pregnant Women and Evaluation of Its Effectiveness: Hatay, Narlıca Sample
Brief Title: Development of Post-Disaster Care Protocol for Pregnant Women and Evaluation of Its Effectiveness
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sakarya University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: E-16214662-050.01.04-284395-97
Record Dates: First submitted 2025-03-10; First posted 2025-07-10 (Actual); Last update posted 2025-07-10 (Actual); Status verified 2025-06

CONDITIONS: Earthquake; Pregnant Women; Support

STUDY DESIGN:
Intervention Model Description: . With this research, the physical and psychosocial needs of pregnant women in the disaster area will be determined. In the second stage, Stevens' Star Model: Transformation of Information model will be used while developing the draft Care Protocol.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- First stage a qualitative and quantitative (parallel design) research was planned (Experimental): In the second stage, Stevens' Star Model: Transformation of Information model will be used while developing the draft Care Protocol.. Necessary permissions have been obtained from Stevens for the use of this model.
  For the applicability and comprehensibility of the care protocol, which was developed as a draft after expert opinions, a pre-application/pilot application will be made with 5-7 pregnant women and the final version will be given. At the end of this stage, a Post-Disaster Care Training Manual for Pregnant Women will be developed. In the third stage, a randomized controlled experimental study will be conducted to determine whether the care protocol to be developed positively affects the physical and psychological health of pregnant women in the disaster area. In line with this goal, 43 pregnant women will be included in the intervention group and 43 pregnant women will be included in the control group.
  Interventions: Behavioral: positively affects the physical and psychological health of pregnant women in the disaster area.

INTERVENTIONS:
Behavioral: positively affects the physical and psychological health of pregnant women in the disaster area. — As time passes after the earthquake, psychological first aid services are not sufficient. Developing a care protocol to provide physical and psychosocial support to pregnant women who are earthquake victims, especially those in the vulnerable group, during the post-disaster disappointment period (months 2-36), is an important unique value of this project.

SUMMARY:
It was designed as a randomized controlled experimental study to determine whether the care protocol planned for pregnant women in the disaster area positively affects their physical and psychological health.

DETAILED DESCRIPTION:
The results of this study suggest that spousal and family support has a positive impact on psychosocial health during pregnancy for women who become pregnant after an earthquake. It was determined that participants had difficulties in accessing health services and exhibited symptoms of fear, sleep disorders, depression and trauma. However, pregnancy, even if unplanned, was considered a hope for a new beginning for many women after a devastating earthquake. The study also emphasizes the importance of pregnant women's need for spiritual care, support and especially attention during this process. In summary, comprehensive mental health support will play a critical role in improving the well-being of earthquake-affected pregnant women.

ELIGIBILITY:
Inclusion Criteria:

* Over the age of 18,
* Positive (+) pregnancy,
* Able to read and write Turkish and speak and understand Turkish,
* No mental or psychological disorder that would cause difficulty in expressing oneself,
* Not receiving a score between 20-27 (severe depression) on HSA-9,
* No chronic disease or high-risk pregnancy diagnosis requiring hospitalization and follow-up,
* Volunteer to participate in the study

Exclusion Criteria:

* Under 18 years of age,
* Foreign nationals who cannot read or write Turkish and are inadequate in speaking or understanding Turkish,
* Those with any mental or psychological disorder/diagnosis,
* Those who score between 20-27 (severe depression) on HSA-9,
* Those with a chronic disease or a diagnosis of high-risk pregnancy requiring hospitalization and follow-up,
* Those who do not agree to participate in the study

Ages: 19 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Estimated)
Dates: Start 2025-03-09 (Actual); Primary Completion 2025-11-15 (Estimated); Study Completion 2026-03-15 (Estimated)

PRIMARY OUTCOMES:
Determining patient health level | The first data will be collected up to the 16th week of pregnancy, the second data between the 36th and 38th weeks, and the last data between the 4th and 8th weeks postpartum.
  PATIENT HEALTH QUESTIONNAIRE - 9 (PHQ-9))
Determining the level of psychosocial health during pregnancy | The first data will be collected up to the 16th week of pregnancy, the second data between the 36th and 38th weeks.
  PSYCHOSOCIAL HEALTH ASSESSMENT SCALE IN PREGNANCY
Determining the level of trauma after an earthquake | The first data will be collected up to the 16th week of pregnancy, the second data between the 36th and 38th weeks, and the last data between the 4th and 8th weeks postpartum.
  POST-EARTHQUAKE TRAUMA LEVEL DETERMINATION SCALE (PSTDBÖ) POST-EARTHQUAKE TRAUMA LEVEL DETERMINATION SCALE (PSTDBÖ)
Determining the level of postpartum depression | The data will be collected between the 4th and 8th weeks postpartum.
  EDINBURG POSTPARTUM DEPRESSION SCALE

CONTACTS AND LOCATIONS:
Overall Officials: Hatice Tambağ, Prof.Dr., Study Director — Hatay Mustafa Kemal Üniversitesi
Locations (1):
- Hatay Mustafa Kemal Üniversitesi, Hatay, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No